CLINICAL TRIAL: NCT02085239
Title: Comparison of Long Acting vs. Short Acting Anesthetic Agents as a Tool for Improving Pain Management Post Ultrasound Guided Breast Biopsy
Brief Title: Comparison of Long vs. Short Acting Anesthesia for Improving Pain Management After Breast Biopsy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never got started; can't delete results
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13027-13-033
Record Dates: First submitted 2014-03-07; First posted 2014-03-12 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2017-04

CONDITIONS: Pain Management After Breast Biopsy
Keywords: Breast Biopsy; Ultrasound; Lidocaine; Ropivacaine; Breast Lesion
MeSH Terms: interventions — Ropivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine alone (Active Comparator): Lidocaine: 8-10 ml of Lidocaine by subcutaneous injection
  Interventions: Drug: Lidocaine alone
- Lidocaine Ropivacaine (Experimental): Lidocaine Ropivacaine
  * 8-10 ml of Lidocaine given by subcutaneous injection
  * 8-10 ml of Ropivacaine given by subcutaneous injection
  Interventions: Drug: Lidocaine Ropivacaine

INTERVENTIONS:
Drug: Lidocaine Ropivacaine — * 8-10 ml of Lidocaine given by subcutaneous injection
  * 8-10 ml of Ropivacaine given by subcutaneous injection
  Other Names: Naropin; Ropivacaine HCL
  Arms: Lidocaine Ropivacaine
Drug: Lidocaine alone
  Arms: Lidocaine alone

SUMMARY:
This study will evaluate the potential role of a long acting anesthetic (ropivacaine) in providing an extended period of pain relief for patients undergoing ultrasound guided core biopsy of the breast.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the potential role of a long acting anesthetic (ropivacaine) in providing an extended period of pain relief for patients undergoing ultrasound guided core biopsy of the breast. One group of patients will receive lidocaine alone for local anesthesia. A second group of patients will similarly receive lidocaine prior to tissue sampling, followed by infiltration of the biopsy area with ropivacaine.

Our hypothesis is that patients who receive a long acting anesthetic (ropivacaine) along with the popular short acting anesthetic (lidocaine), will be pain free after the breast biopsy procedure for a longer period of time than the patients who only receive lidocaine (the short acting anesthetic). This will lessen the emotional and physical trauma associated with the procedure and give patients a better experience thereby improving patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast lesions recommended for biopsy by physician

Exclusion Criteria:

* Patients with breast lesions not recommended for biopsy
* Patients with allergic reactions to lidocaine, ropivacaine, or related anesthetics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in pain level from baseline to 1 hour | 1 hour after procedure
  Amount of pain that patient is feeling at baseline and 1 hour after the procedure

SECONDARY OUTCOMES:
Change in pain level from 1 hour to 5 hours after procedure | 5 hours
  Amount of pain that patient is feeling 5 hours after the procedure
Change in pain level from 5 to 10 hours after the procedure | 10 hours after procedure
  Amount of pain that patient is feeling 10 hours after the procedure
Change in pain level from 10 to 24 hours after procedure | 24 hours after procedure
  Amount of pain that patient is feeling 24 hours after the procedure
Pathology | up to 72 hours after procedure
  Description of tissue collected Benign or malignant tumor (if found) Type of tumor

CONTACTS AND LOCATIONS:
Overall Officials: Dean Shanley, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Mary Jo Cropper Family Center for Breast Care; Bethesda North Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Applied Radiology. Breast biopsy: Anesthesia, bleeding prevention, representative sampling and rad-path concordance. Vol 41.1. Jan 2012
- [Background] Reynolds HE, Jackson VP, Musick BS. Preoperative needle localization in the breast: utility of local anesthesia. Radiology. 1993 May;187(2):503-5. doi: 10.1148/radiology.187.2.8475298.
- [Background] Novy DM, Price M, Huynh PT, Schuetz A. Percutaneous core biopsy of the breast: correlates of anxiety. Acad Radiol. 2001 Jun;8(6):467-72. doi: 10.1016/S1076-6332(03)80617-7. PMID 11394538